CLINICAL TRIAL: NCT01421875
Title: Genetic and Epigenetic Determinants of Chemotherapy Resistance and Adverse Outcome in Elderly Patients With AML
Brief Title: Biomarker Study of Chemotherapy Resistance and Outcomes in Samples From Older Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000709403; ECOG-E3999T4
Record Dates: First submitted 2011-08-20; First posted 2011-08-23 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with del(5q); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); untreated adult acute myeloid leukemia; adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); adult acute megakaryoblastic leukemia (M7); adult acute minimally differentiated myeloid leukemia (M0)
MeSH Terms: conditions — Leukemia; Congenital Abnormalities; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute | interventions — DNA Methylation; Gene Expression Profiling; Microarray Analysis; Base Sequence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Genetic: DNA methylation analysis
Genetic: RNA analysis
Genetic: gene expression analysis
Genetic: microarray analysis
Genetic: nucleic acid sequencing
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying blood samples from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research trial studies biomarkers related to chemotherapy resistance and outcomes in samples from older patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Delineate the spectrum of genetic and epigenetic lesions occurring in elderly patients with acute myeloid leukemia (AML).
* Determine the biological functions perturbed by these lesions.
* Identify and validate lesions or pathways that are most highly associated with chemo-sensitive and chemo-refractory disease, and with adverse outcome in elderly AML.
* Identify potential classifiers and biomarker lesions that we can then evaluate prospectively in the E2906 trial which is about to begin enrollment.

OUTLINE: DNA and RNA extracted from cell samples are analyzed for genetic and epigenetic expression by Agilent SureSelect sequencing, Illumina HiSeq2000 platform coding and sequencing, DNA methylation, and microarray assays. Results are then associated with patients' overall survival, progression-free survival, and complete response rate. Results are also analyzed assessing the prognostic relevance of known mutations and epigenetic alterations that have shown to have an impact on overall survival and response to therapy in younger patients with acute myeloid leukemia (AML) in E1900 including, but not limited to, FLT3, DNMT3A, IDH1, IDH2, TET2, ASXL1, WT1, and MLL, and 15-gene DNA methylation classifier, and with novel recurrent mutations identified by other AML-profiling efforts.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Subset of patients diagnosed with acute myeloid leukemia (AML) enrolled on E3999
* AML resistant or sensitive to chemotherapy
* Mononuclear cell samples available

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 61 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples from patients enrolled E3999 from whom samples were submitted for research
Sampling Method: Non-Probability Sample
Enrollment: 257 (Actual)
Dates: Start 2011-08-17 (Actual); Primary Completion 2011-10-17 (Actual); Study Completion 2011-10-17 (Actual)

PRIMARY OUTCOMES:
Genetic and epigenetic determinants of chemoresistance and adverse outcomes | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ross Levine, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center